CLINICAL TRIAL: NCT01065805
Title: A Contiguous, Sequential Phase I/II Imaging Study of 18F-fluoro-3'-L-fluorothymidine (18F-FLT) in Patients With Known or Suspected Carcinoma of the Lung, Breast, Renal Cell, Pancreas, or Brain, and With Gastrointestinal Malignancies, Neuroendocrine Tumours or Lymphoma
Brief Title: A Study to Demonstrate the Safety and Preliminary Efficacy of 18F-FLT in Patients With Solid Tumours or Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Retirement of former Qualified Investigator and lack of resources to complete study
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-FLT-002
Record Dates: First submitted 2008-12-19; First posted 2010-02-09 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-02

CONDITIONS: Brain Cancer; Cancer; Solid Tumor; Lymphoma
Keywords: 18F-FLT; Positive Emission Tomography; Cancer
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Lymphoma | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18F-FLT PET
  Interventions: Biological: 18F-FLT

INTERVENTIONS:
Biological: 18F-FLT — Phase I: Radioactive dose of 2.59 MBq/kg (111-222 MGq)per injection. A single injection of 18F-FLT and PET scan will be permitted per patient.
  Phase II: Radioactive dose of 2.59 MBq/kg (100-350) MBq per injection. Up to five separate injections of 18F-FLT and PET scans will be permitted per patient

SUMMARY:
The Radiotracer 18F-FLT can non-invasively assess excessive cell growth in PET scan images. Tumour growth rate is a useful indicator of tumour aggression and response to treatment. Imaging and measuring the cell growth with 18F-FLT may be useful in monitoring response to anticancer treatment.

DETAILED DESCRIPTION:
Clinical trial is a combined Phase I/II imaging, open label, single site study in patients with known or suspected carcinoma of the lung, breast, renal cell, pancreas or brain, and with gastrointestinal malignancies, neuroendocrine tumours, or lymphoma. One 18F-FLT PET scan will be performed in 10 Phase I patients, and pre-injection and post-imaging blood work and vital signs will be collected. Up to 5 18F-FLT PET scans will be performed in 170 Phase II patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 16 years of age. If female of child-bearing potential and outside of the window of 10 days since the first day of last menstrual period, a negative pregnancy test is required.
* Patients with known primary or suspected primary, recurrent or metastatic carcinoma of the lung, breast, renal cell, pancreas or brain (including GGM, oligodendrogliomas, and brain metastases from any primary tumour) and with gastrointestinal malignancies, neuroendocrine tumours (including carcinoid and islet cell malignancies, or lymphoma, with at least one lesion >1 cm in diameter.
* Biochemical parameters as measured are required to be within 5 times the normal limits for age.
* Able and willing to follow instruction and comply with the protocol
* Provide written informed consent prior to participation in the study
* Karnofsky Performance Scale Score 50-100

Exclusion Criteria:

* Previous removal of entire tumour
* Biochemical parameters as measured outside 5 times the normal limits for age
* Unable or unwilling to follow instructions and comply with the protocol
* Unable or unwilling to provide written informed consent prior to participation in the study
* Karnofsky Performance Scale Score < 50
* Nursing or pregnant females
* Age less than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-03-20 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Phase I: to determine the safety of 18 F-FLT. | 3 years
Phase II: To determine general biodistribution of 18F-FLT and correlate 18F-FLT uptake with hENT1 expression and Ki-67 scores. | 3 years

SECONDARY OUTCOMES:
Phase I: To determine general biodistribution of 19F-FLT | 3 years
Phase II: to confirm safety of 18F-FLT; to determine the relative uptake of 18F-FLT (SUV, RUS, T/N); and to correlate 18F-FLT uptake with patient outcomes. | 3 years
Phase II: to correlate 18F-FLT uptake with patient outcomes (treatment response, progression-free survival, overall survival), over the first 12 months of follow-up after completion of tx, subsequently over the remainder of the disease course | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sawyer, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada